CLINICAL TRIAL: NCT03124121
Title: Study of the Golimumab Exposure-Response Relationship Using Serum Trough Levels
Acronym: GO-LEVEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-001374-42
Record Dates: First submitted 2017-04-04; First posted 2017-04-21 (Actual); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Induction cohort (Other): Golimumab induction therapy
  Interventions: Drug: Golimumab
- Maintenance cohort (Other): Golimumab maintenance therapy
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Golimumab — A biologic agent which acts by antagonising the effects of tumour necrosis factor (TNF) alpha
  Other Names: Simponi

SUMMARY:
The purpose of this study is to gain insight into the exposure-response relationship of golimumab in moderate-to-severe Ulcerative Colitis (UC).

Patients commencing induction therapy with golimumab will be enrolled into a prospective study and evaluated at three time-points (weeks 6, 10 and 14) for clinical and biochemical UC disease activity as well as serum golimumab concentrations and the presence of anti-golimumab antibodies. Patients already established on stable golimumab maintenance therapy will be enrolled into a cross-sectional study with the same evaluations taken at a single time point.

DETAILED DESCRIPTION:
The study will involve two study groups designed to offer insights into the pharmacokinetics of golimumab during induction and maintenance therapy:

Cohort 1: Patients commencing golimumab induction therapy will be included in a prospective, observational study.

Cohort 2: Patients receiving golimumab maintenance therapy will be included in a cross-sectional, observational study.

Primary objective: To define a week 6 serum golimumab concentration that predicts response at week 14.

Secondary objective: To define serum golimumab concentrations at weeks 6, 10 and 14 that predict response at each time point, respectively and at week 14.

Exploratory objectives:

Correlations between serum golimumab concentrations and novel disease activity indices (PRO2), biochemical markers of disease activity (CRP, faecal calprotectin) and quality of life indices (IBD-Q and IBD-Control).

Correlations between the presence of anti-golimumab antibodies, serum golimumab concentrations and UC disease activity.

This study will also generate data that can be used to validate a commercially available golimumab assay as well as a novel patient reported outcome (PRO) assessment of clinical UC disease activity.

ELIGIBILITY:
Inclusion Criteria for cohort 1:

* Aged 18 years or over
* Moderate-to-severe UC, defined as:

SCCAI > 5 and, i. A raised fecal calprotectin (> 59 μg/g) or, ii. A raised CRP (> 5 mg/L) or, iii. Endoscopic disease activity Mayo 2 or above, Evaluated within 4 weeks of study enrollment

* Commencing golimumab treatment
* Written informed consent to participate
* Sufficient English language skills to understand the patient information sheet and consent form

Inclusion Criteria for cohort 2:

* Aged 18 years or over
* Receiving golimumab treatment for UC for over 18 weeks (6 injections)
* Written informed consent to participate
* Sufficient English language skills to understand the patient information sheet and consent form

Exclusion Criteria (cohort 1 only):

* Contra-indication to golimumab: tuberculosis or severe infections
* Imminent need for colectomy (i.e. colectomy is being planned)
* Previous primary non-response to anti-TNF therapy in the opinion of the investigator
* Previous treatment with more than one anti-TNF therapy (excluding golimumab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samaan MA, Cunningham G, Tamilarasan AG, Beltran L, Pavlidis P, Ray S, Mawdsley J, Anderson SH, Sanderson JD, Arkir Z, Irving PM. Therapeutic thresholds for golimumab serum concentrations during induction and maintenance therapy in ulcerative colitis: results from the GO-LEVEL study. Aliment Pharmacol Ther. 2020 Jul;52(2):292-302. doi: 10.1111/apt.15808. Epub 2020 Jun 7. PMID 32506695

RESULTS

PARTICIPANT FLOW:
Groups:
- Golimumab Induction Therapy: Patients commencing golimumab
- Golimumab Maintenance Therapy: Patients receiving golimumab maintenance therapy
Period: Overall Study
Arm/Group | Golimumab Induction Therapy | Golimumab Maintenance Therapy
Started | 42 | 70
Completed | 39 | 67
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Golimumab Induction Therapy | Golimumab Maintenance Therapy | Total
Number analyzed (Participants) | 39 | 67 | 106
Age, Continuous [Median (Full Range); unit: years] | 37 [24 to 48] | 36 [20 to 73] | 36 [20 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 30 | 47
  Male | 22 | 37 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Serum Golimumab Concentration (μg/ml)
Description: Evaluated using an enzyme-linked immunosorbent assay (ELISA)
Time Frame: Week 6 during induction therapy and at the point of study entry during maintenance
Measure: Median (Full Range); unit: ug/ml
Arm/Group | Golimumab Induction Therapy | Golimumab Maintenance Therapy
Number analyzed (Participants) | 39 | 67
ug/ml | 3.3 [1.3 to 8.0] | 2.4 [0.6 to 7.4]

2. Secondary Outcome: Number of Patients in Clinical Remission
Description: Evaluated using the Simple Clinical Colitis Activity Index (SCCAI). Remission defined as SCCAI < 3.
Time Frame: Week 14 during induction therapy and at the point of study entry during maintenance therapy
Measure: Count of Participants; unit: Participants
Groups:
- Induction Cohort: Patients commencing golimumab
- Maintenance Cohort: Patients receiving golimumab maintenance therapy
Arm/Group | Induction Cohort | Maintenance Cohort
Number analyzed (Participants) | 42 | 67
Participants | 22 | 41

3. Secondary Outcome: Faecal Calprotectin (μg/g)
Description: Faecal inflammatory marker with higher values suggestive of increasing biochemical disease activity
Time Frame: Week 14 during induction therapy and at the point of study entry during maintenance
Measure: Median (Full Range); unit: ug/g
Arm/Group | Golimumab Induction Therapy | Golimumab Maintenance Therapy
Number analyzed (Participants) | 42 | 63
ug/g | 46 [5 to 2000] | 57 [5 to 1260]

4. Secondary Outcome: Serum C-Reactive Protein (mg/L)
Description: Serum inflammatory marker with higher values suggestive of increasing biochemical disease activity
Time Frame: Week 14 during induction therapy and at the point of study entry during maintenance
Measure: Median (Full Range); unit: mg/L
Arm/Group | Golimumab Induction Therapy | Golimumab Maintenance Therapy
Number analyzed (Participants) | 42 | 67
mg/L | 1 [1 to 50] | 1 [1 to 21]

5. Secondary Outcome: Serum Albumin (g/L)
Description: Serum protein marker with higher values associated with increasing inflammatory activity and lower serum levels of anti-TNF agents (such as golimumab)
Time Frame: Week 14 during induction therapy and at the point of study entry during maintenance
Measure: Median (Full Range); unit: g/L
Arm/Group | Golimumab Induction Therapy | Golimumab Maintenance Therapy
Number analyzed (Participants) | 42 | 67
g/L | 46 [33 to 52] | 47 [40 to 54]

6. Secondary Outcome: Clinical UC Disease Activity
Description: Evaluated using Patient Reported Outcome 2 (PRO2). PRO2 ranges from 0-5 with higher scores denoting increasing clinical disease activity.
Time Frame: Week 14 during maintenance therapy and at the point of study entry during maintenance
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Golimumab Induction Therapy | Golimumab Maintenance Therapy
Number analyzed (Participants) | 42 | 67
score on a scale | 1 [0 to 5] | 0 [0 to 5]

7. Secondary Outcome: Quality of Life (IBD-Control)
Description: Evaluated using IBD-Control questionnaires. IBD-Control scores range from 0-16 with higher scores denoting better quality of life.
Time Frame: Week 14 during induction therapy and at the point of study entry during maintenance therapy
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Golimumab Induction Therapy | Golimumab Maintenance Therapy
Number analyzed (Participants) | 42 | 67
score on a scale | 12.5 [0 to 16] | 14 [0 to 16]

8. Secondary Outcome: Number of Patients With Detectable Anti-golimumab Antibodies
Description: Evaluated using a drug-sensitive enzyme-linked immunosorbent assay (ELISA)
Time Frame: At any study time point during induction therapy (weeks 6, 10 or 14) and at the point if study entry during maintenance
Measure: Count of Participants; unit: Participants
Arm/Group | Golimumab Induction Therapy | Golimumab Maintenance Therapy
Number analyzed (Participants) | 42 | 67
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: During the 14 week induction study for patients commencing treatment and at a single time point (the point of recruitment) for patients on maintenance therapy.
Description: Only serious adverse events (including all-cause mortality) were recorded. Non-serious adverse events were not recorded.
Groups:
- Golimumab Induction Therapy: Patients commencing golimumab induction
Arm/Group | Golimumab Induction Therapy | Golimumab Maintenance Therapy
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/70
Serious Adverse Events (participants affected / at risk) | 4/42 | 0/70
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Golimumab Induction Therapy (N=42) | Golimumab Maintenance Therapy (N=70)
Facet join injection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) — Azathioprine induced pancreatitis
Ulcerative colitis flare requiring admission (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT03124121/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03124121/ICF_001.pdf